CLINICAL TRIAL: NCT01556893
Title: Prospective, Single-center Clinical Trial of Subjects Scheduled to Undergo LASIK Surgery Requiring an Initial Corneal Flap.
Brief Title: Creating LASIK Flaps With the LenSx Femtosecond Laser
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon LenSx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-004f
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Myopia; Hyperopia
Keywords: Flap Creation; Femtosecond Laser; corneal flap prior to LASIK procedure
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LASIK Flap Arm (Other): This is a single arm study.
  Interventions: Device: LenSx Laser

INTERVENTIONS:
Device: LenSx Laser — The LenSx laser system is a femtosecond laser that has received 510(k) clearance for anterior capsulotomy during cataract surgery (K082947), laser phacofragmentation during cataract surgery (K094052) and for use in the creation of a single and multi-plane arc cut/incisions in the cornea (K092647).

SUMMARY:
This will be a prospective, single-center clinical trial of up to 50 eyes of subjects scheduled to undergo LASIK surgery requiring an initial corneal flap. Subjects will be screened for eligibility.

Subjects will undergo LASIK surgery using the LenSx Laser to create the corneal flap prior to excimer laser treatment.

Subjects will be evaluated intraoperatively to assess the ease of lifting the flaps, the stromal bed quality, and the amount of opaque bubble layer. All patients will be followed with routine vision exams for 3 months postoperatively to evaluate changes in visual acuity, manifest refraction, slit lamp examination, and endothelial cell counts.

ELIGIBILITY:
Inclusion Criteria:

1. Must have myopia or hyperopia eligible for femtosecond initiated LASIK surgery
2. Must be over 18 years of age
3. Must have visual acuity correctable to at least 20/25 in both eyes
4. If subject is a contact lens wearer, discontinuation of contact lens wear prior to preoperative exam (2 weeks prior for soft contact lenses, 4 weeks prior for rigid gas permeable contact lenses, and 8 weeks prior for hard contact lenses)
5. Must be willing and able to return for scheduled follow up examinations through 3 months after surgery
6. Must sign and be given a copy of the written Informed Consent form
7. Postoperative refractive target is emmetropia

Exclusion Criteria:

1. Known sensitivity to planned study concomitant medications
2. Participation in any other ophthalmic drug or device clinical trial during the time of this clinical investigation
3. Presenting any contraindications to femtosecond initiated LASIK
4. Corneal thickness values that will result in residual bed less than 280 microns when flap resection and excimer ablation are calculated
5. Irregular astigmatism, based on Investigator's judgment
6. Undergoing monovision LASIK
7. Pregnant, lactating or plan to become pregnant during the course of this study
8. For bilateral second study eyes only: The surgeon shall not proceed with the second eye until the 1 week exam of the first eye shows no vision threatening complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Ease of Lifting Flaps | Operative
  0 - Unable to lift flap
  1. - Able to lift flap with aid of sharp instrument
  2. - Able to lift flap with difficulty using blunt instrument
  3. - Able to lift flap with moderate resistance using blunt instrument
  4. - Able to lift flap with minimal resistance using blunt instrument
  5. - Able to lift flap without any resistance using blunt instrument (Scale)

SECONDARY OUTCOMES:
Stromal Bed Quality | Operative
  0 - very rough
  1- moderately rough 2 - rough 3 - smooth 4 - moderately smooth 5 - very smooth (Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Semmelweis University, Budapest, Hungary